CLINICAL TRIAL: NCT00715169
Title: Phase 2 A, Double-Blind, Randomized, Placebo-Controlled Trial Measuring the Effects of MLN1202 on C-Reactive Protein Levels in Patients With Risk Factors for Cardiovascular Disease
Brief Title: Double-Blind, Randomized, Placebo-Controlled Trial of MLN1202 on C-Reactive Protein Levels in Patients With Risk Factors for Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Clinical Research Monitor, Millennium Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN1202
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — plozalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: MLN1202
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MLN1202 — 10 mg/kg dose of MLN1202 administered via IV infusion administered approximately 30 minutes to an hour
  Arms: 1
Other: Placebo — Placebo consist of 0.9% saline solution administered as a 10 mg/kg dose via IV infusion administered approximately 30 minutes to an hour
  Arms: 2

SUMMARY:
This study is a, randomized, double-blind, placebo-controlled phase 2a trial evaluating the potential of MLN1202 to reduce circulating levels of C-reactive protein (CRP)in patients with risk factors for Atherosclerotic cardiovascular disease (ASCVD). Patients with risk factors for ASCVD will be screened for inclusion and exclusion criteria including assessment of C-reactive protein. If the patient's CRP is greater than 3.0 mg/L on repeated measurements at least 2 weeks apart, the patient will be enrolled, stratified by screening CRP levels (≤5.0 mg/L and >5.0 mg/L), and randomized to receive 1 dose of either placebo or MLN1202. Safety will be assessed by vital signs, physical examination, clinical laboratories at baseline, and adverse event (AE) reporting from Day 1 to Day 113 of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 35 years or older
* Willing and able to comply with the protocol for the duration of the study
* Willing to use adequate double-barrier contraceptive methods for the duration of the study
* Presence of 2 or more of the following risk factors for ASCVD:

Age of 45 years (male) or 55 years (female) or greater History of or current cigarette smoking of ≥20 pack years History of hypertension Body mass index (BMI) defined as weight (kg) divided by height (in m2) ≥30 History of hypercholesterolemia defined as fasting low-density lipoprotein >130 mg/dL History of high-density lipoprotein levels of 40 mg/dL or less Diabetes mellitus Family history of a definable ASCVD event (myocardial infarction or intervention)in a first-degree relative prior to the age of 55 (male) or 65 (female)

* Patients with hypercholesterolemia may be on stable doses of lipid-lowering agents with no change in regimen/dose within 60 days prior to randomization
* Have high-sensitivity C-reactive protein (from peripheral blood) levels >3.0 mg/L on more than 1 test date separated by at least 2 weeks in the last 12 months; the most recent hsCRP must be measured during Screening within 14 days of randomization

Exclusion Criteria:

* History of stroke History of acute coronary syndrome (ACS) including unstable angina, acute myocardial infarction (both ST segment elevation and non-ST segment elevation) or stable angina
* Evidence of coronary artery disease as determined by either prior history of CAD-related event (stable angina, unstable angina, MI) or evidence on diagnostic procedure (exercise stress test, echocardiogram, stress test, radionucleotide stress test, others) that in the opinion of the investigator is consistent with CAD
* Diagnosis of congestive heart failure or clinical evidence suggesting CHF including history of orthopnea, exertional dyspnea, pedal edema, pulmonary rales, hepatosplenomegaly, cardiomegaly, and a prediastolic (S3) gallop
* Uncontrolled hypertension with a blood pressure >140/90 at Screening
* Concurrent chronic inflammatory illness (eg, inflammatory bowel disease, rheumatoid arthritis, chronic obstructive pulmonary disease, asthma, systemic lupus erythematosus) or concurrent chronic infectious illness (eg, human immunodeficiency virus, tuberculosis, hepatitis, osteomyelitis)
* Concurrent use of anti-inflammatory or disease-modifying agents (eg, methotrexate,azathioprine, oral corticosteroids). Past use (>3 months) of these anti-inflammatory ordisease modifying agents is acceptable. Aspirin, clopidogrel, and nonsteroidal antiinflammatory drugs are acceptable
* History of cancer with the exception of cervical carcinoma-in-situ or basal cell carcinoma of the skin within the last 5 years
* History of receiving live attenuated vaccine within last 60 days prior to randomization
* Use of an investigational product in the last 60 days prior to randomization
* History of illicit drug use or alcohol abuse in the last year
* History of or planned percutaneous coronary intervention, such as angioplasty or coronary stent placement, or coronary artery bypass graft or other vascular surgery planned within study duration
* Chest X-ray within 6 months prior to study entry with clinically significant findings, in the opinion of the investigator Screening electrocardiogram obtained once during Screening Days -14 to -1 with clinically significant findings, in the opinion of the investigator
* Renal function reflected by a serum creatinine ≥1.5 times the upper limit of normal
* Hepatic function reflected by elevated liver function tests (eg, aspartate aminotransferase, alanine aminotransferase or total bilirubin) ≥2 times the ULN
* If female, positive results on a serum pregnancy test or breastfeeding
* Any other reason in the opinion of the investigator that a subject should not be enrolled in this study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of C-C Chemokine Receptor-2 (CCR2) blockade in reducing Creactive protein (CRP) levels in patients with risk factors for atherosclerotic cardiovascular disease (ASCVD) and a baseline elevation of CRP | The change from baseline to Day 57 in CRP between patients treated withplacebo compared with MLN1202

SECONDARY OUTCOMES:
Elevation of Creactive protein (CRP) number of days from baseline until the first 1.0 mg/L decrease in CRP levels and changes from baseline to other study visits. | Baseline, Day 1 to Day 113 of the trial.